CLINICAL TRIAL: NCT01547663
Title: A Comparison of Pain Scales in Patients With Disorder of Consciousness Following Craniotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwannee Suraseranivongse, Professor, Mahidol University
Other Study IDs: SIRB 461/2554
Record Dates: First submitted 2012-03-04; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Pain, Postoperative
Keywords: pain scale; craniotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to test validity, reliability and practicality of translated NCS, CNPI and FLACC in unconscious patients in 48 hour following craniotomy.

DETAILED DESCRIPTION:
This study aims to test predictive validity (sensitivity and specificity), content validity, concurrent validity, construct validity, inter-rater reliability and practicality of translated Nociception Coma Scale (NCS) , Checklist of Non Verbal Pain Indicator (CNPI) and the Faces, Legs, Activity, Cry, Consolability Observation Tool (FLACC) in unconscious patients in 48 hour following craniotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Preoperative intracranial lesion which predicts delayed recovery
3. Disorder of consciousness within 48 hours after craniotomy assessed by using Coma Recovery Scale-Revised (CRS-R) 17
4. Not received postoperative sedation or muscle relaxants

Exclusion Criteria:

1. Documented history of prior brain injury
2. History of delayed development
3. Prior psychiatric illness
4. Prior neurological illness
5. Superior limb contusion, fracture, paralysis -cannot move
6. Thalamic hemorrhage -cannot express feeling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with disorder of consciousness within 48 hours following craniotomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand